CLINICAL TRIAL: NCT01805232
Title: Intravenous Artesunate Versus Quinine in Severe Malaria at Kassla, Sudan
Brief Title: Intravenous Artesunate and Malaria
Acronym: IVAS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Khartoum (Other)
Collaborators: University of Kassala, Sudan (Other); Kassala (Unknown); Sudan (Unknown)
Responsible Party: Principal Investigator, Ishag Adam, Professor, University of Khartoum
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: artesunate and malaria
Record Dates: First submitted 2013-03-02; First posted 2013-03-06 (Estimated); Last update posted 2013-03-06 (Estimated); Status verified 2013-03

CONDITIONS: Malaria
Keywords: severe; Falciaparum; Malaria
MeSH Terms: conditions — Malaria; Lymphoma, Follicular | interventions — Artesunate; Quinine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- artesunate (Experimental): intravenous artesunate 80 mg/kg initially then after 8 hours then daily
  Interventions: Drug: artesunate; Drug: Quinine
- quinine (Active Comparator): quinine infusion 80 mg/kg every 8 hours
  Interventions: Drug: artesunate; Drug: Quinine

INTERVENTIONS:
Drug: artesunate — intravenous artesunate 80 mg/kg initially then after 8 hours then daily
Drug: Quinine — quinine infusion 80 mg/kg every 8 hours till the patient can take orally

SUMMARY:
Intravenous artesunate is egual to quinine in the treatment of severe malaria

DETAILED DESCRIPTION:
Intravenous artesunate is egual to quinine in the treatment of severe malaria in the form of fever clearance time and parasite clearance time

ELIGIBILITY:
Inclusion Criteria:

severe P.falciparum malaria-

Exclusion Criteria:

mixed infection Pregnant women -

Ages: 1 Year to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2013-03; Primary Completion 2013-05 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
clearance of the parasite and fever | 3 days
  To compare the parasite clearance time and fever clearance time between the two groups

CONTACTS AND LOCATIONS:
Locations (1):
- Kassala, Kassala, Kassala, Sudan

REFERENCES:
- [Background] Eltahir HG, Omer AA, Mohamed AA, Adam I. Comparison of artesunate and quinine in the treatment of Sudanese children with severe Plasmodium falciparum malaria. Trans R Soc Trop Med Hyg. 2010 Oct;104(10):684-6. doi: 10.1016/j.trstmh.2010.05.009. Epub 2010 Jun 17. PMID 20850004